CLINICAL TRIAL: NCT01527682
Title: Efficacy and Safety of Prostaglandin Analogue and Carbonic Anhydrase Inhibitor for the Treatment of Pediatric Glaucoma
Brief Title: Efficacy and Safety of Topically Applied Medical Therapy for the Treatment of Pediatric Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Luciano Quaranta MD, Associate Professor in Ophthalmology, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-004763-19
Record Dates: First submitted 2010-02-16; First posted 2012-02-07 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Childhood Glaucoma
Keywords: Intraocular pressure; Latanoprost; Dorzolamide
MeSH Terms: conditions — Hydrophthalmos | interventions — Latanoprost; dorzolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Latanoprost, Dorzolamide (Other): According to intraocular (IOP) assessment, the eye will receive Latanoprost, Dorzolamide or both.
  Interventions: Drug: Latanoprost, Dorzolamide

INTERVENTIONS:
Drug: Latanoprost, Dorzolamide — * Latanoprost 0.005% ophthalmic solution given once a day at nighttime (9.00 PM)
  * Dorzolamide 2% ophthalmic solution given three times a day as a monotherapy, two times a day if in combination with latanoprost
  Other Names: - Latanoprost, a prostaglandin analogue; - Dorzolamide, a potent inhibitor of carbonic anhydrase II

SUMMARY:
Objectives:

The study will assess the ocular hypotensive effect of latanoprost and dorzolamide in a selected sample of patients affected by primary Pediatric Glaucoma (PG), refractory to surgical procedures. Safety will be assessed, too.In the first version of the protocol 96 eyes were forecasted to complete the enrolment. The protocol was then amended and now to complete the study 68 eyes should be included. This number of eyes could be achieved by recruiting from 34 to 68 patients due to not in all patients both eyes should be eligible for the study.

DETAILED DESCRIPTION:
Study design:

Single arm, prospective, experimental study. Due to ethical reasons and in order to adhere as much as possible to current clinical practice, the presence of a control arm is not planned. Due to the non-comparative nature of the study, no blinding of treatment is planned.

ELIGIBILITY:
Inclusion Criteria:

* Children of either sexes, aged 0-12 years
* Diagnosis of mono- or bilateral primary congenital glaucoma
* IOP greater than or equal to 22 mmHg and lower than 27 mmHg
* Only one previous ocular hypotensive surgical procedure for treatment of glaucoma among the following: goniotomy, trabeculotomy, trabeculotomy with adjunct of mitomycin C) (only for medical treatment at least one month before)
* Parent informed consent to data processing (at registration)
* Parent informed consent before any study procedure

Exclusion Criteria:

* Secondary glaucoma (Sturge-Weber syndrome, type I neurofibromatosis, retinoblastoma, steroid-induced glaucoma, etc.)
* Presence of concomitant abnormalities of the anterior segment of the eye (cataract, iridocorneal dysgenesia, congenital uveal ectropion uvea, etc.)
* Previous treatment with the study drugs
* Presence of concomitant systemic diseases (asthma, hypertension, cardiac disease, renal failure, etc.) that needs treatment with drugs, that could influence IOP (steroids, beta-blockers, angiotensin-converting-enzyme inhibitor -inhibitors diuretics, etc.)
* Abnormalities of the cornea that could influence IOP readings (marked cornea edema)

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Quaranta, MD, Principal Investigator — Università di Brescia, Spedali Civili di Brescia
Locations (2):
- Italy (2):
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - A.O. Universitaria " Policlinico Vittorio Emanuele" P.O. Rodolico, Catania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uva MG, Avitabile T, Reibaldi M, Bucolo C, Drago F, Quaranta L, Lionetti E, Longo A. Long-term efficacy of latanoprost in primary congenital glaucoma. Eye (Lond). 2014 Jan;28(1):53-7. doi: 10.1038/eye.2013.232. Epub 2013 Oct 25. PMID 24158022
- [Result] Quaranta L, Biagioli E, Galli F, Poli D, Rulli E, Riva I, Hollander L, Katsanos A, Longo A, Uva MG, Torri V, Weinreb RN. Latanoprost and Dorzolamide for the Treatment of Pediatric Glaucoma: The Glaucoma Italian Pediatric Study (Gipsy), Design and Baseline Characteristics. Adv Ther. 2016 Aug;33(8):1305-15. doi: 10.1007/s12325-016-0358-x. Epub 2016 Jun 16. PMID 27312975
- [Result] Quaranta L, Biagioli E, Riva I, Galli F, Poli D, Rulli E, Katsanos A, Longo A, Uva MG, Torri V, Weinreb RN. The Glaucoma Italian Pediatric Study (GIPSy): 1-Year Results. J Glaucoma. 2017 Nov;26(11):987-994. doi: 10.1097/IJG.0000000000000773. PMID 28957960

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive Primary Congenital Glaucoma not sufficiently responder to a single surgical procedure
Pre-assignment Details: Patients affected with Primary congenital glaucoma will be recruited if after a single surgical procedure Intraocular pressure will be ranging from 22 and 27 mm Hg
Units Other Than Participants: eyes
Groups:
- Latanoprost, Dorzolamide: According to IOP assessment, the eye will receive Latanoprost, Dorzolamide or both.
  Latanoprost, Dorzolamide: - Latanoprost 0.005% ophthalmic solution given once a day at nighttime (9.00 PM)
  - Dorzolamide 2% ophthalmic solution given three times a day as a monotherapy, two times a day if in combination with latanoprost
Period: Overall Study
Arm/Group | Latanoprost, Dorzolamide
Started | 37; 69 eyes
Completed | 29; 45 eyes
Not Completed | 8; 24 eyes
Not completed — Protocol Violation | 8

BASELINE CHARACTERISTICS:
Arm/Group | Latanoprost, Dorzolamide
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.1 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 22
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Response
Description: defined as those eyes in which the decrease of intraocular pressure (IOP) of at least 20% with respect to baseline assessment will be achieved and maintained during the 3-year period of study duration
Time Frame: 3 years
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Latanoprost, Dorzolamide
Number analyzed (Participants) | 27
Number analyzed (eyes) | 43
eyes | 33
Statistical Analysis 1: Comparison: Latanoprost, Dorzolamide; Test type: Other; Proportion = 76.7, 95% CI 2-sided [64.1 to 89.4]; The statistical analysis was performed according to study design. Using a Fleming single stage design (A'Hern approach) setting the probability of erroneously concluding that the responders rate is greater than 35% at 5% (one-sided alpha=0.05) and the probability of correctly concluding that the responders rate is at least 50% at 80% (beta error = 0.20), the minimum number of responder eyes was set at 31 out of 68, since this result is associated with a lower limit of the 90% exact confidence interval of 35.2%

2. Secondary Outcome: Time to Treatment Failure (TTF)
Description: calculated as the time from the date of baseline visit to the date in which the medical treatment will be stopped, since IOP control will be considered not satisfactory
Time Frame: 3 years
Measure: Median (Inter-Quartile Range); unit: eyes
Units Other Than Participants: eyes
Arm/Group | Latanoprost, Dorzolamide
Number analyzed (Participants) | 29
Number analyzed (eyes) | 45
eyes | NA [NA to NA] — insufficient number of participants with events

3. Secondary Outcome: Number of Eyes With an Adverse Event (AE)
Description: The occurrence of the following events will be monitored: growth of the eyelashes (hypertrichosis), changes iris colour, corneal epitheliopathy, allergic conjunctivitis, increase of central corneal thickness, non-serious and serious adverse event occurrence.
Time Frame: 3 years
Population: Eyes affected by Primary congenital glaucoma not sufficiently responder to a single surgical procedure
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Latanoprost, Dorzolamide
Number analyzed (Participants) | 37
Number analyzed (eyes) | 61
eyes | 61

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Latanoprost / Dorzolamide: According to IOP assessment, the eye will receive Latanoprost, Dorzolamide or both.
  Latanoprost, Dorzolamide: - Latanoprost 0.005% ophthalmic solution given once a day at nighttime (9.00 PM)
  - Dorzolamide 2% ophthalmic solution given three times a day as a monotherapy, two times a day if in combination with latanoprost
Arm/Group | Latanoprost / Dorzolamide
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 22/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Latanoprost / Dorzolamide (N=37)
Hypertrichosis (Eye disorders) | 17
Iris color modification (Eye disorders) | 6
Corneal epitheliopathy (Eye disorders) | 17
Allergic conjunctivitis (Eye disorders) | 9
Eyelid skin hyperpigmentation (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No